CLINICAL TRIAL: NCT04952493
Title: The Efficacy and Safety of Anlotinib Hydrochloride or Penpulimab In Combination With RAI in Patients With Local Advanced or Metastatic Differentiated Thyroid Cancer: A Randomized, Open-label, Exploratory Clinical Trial
Brief Title: Anlotinib or Penpulimab in Combination With RAI for DTC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yansong Lin, Prof. M.D., Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-T002
Record Dates: First submitted 2021-06-27; First posted 2021-07-07 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2021-08

CONDITIONS: Thyroid Cancer
Keywords: Anlotinib; Iodine
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Iodine-131; penpulimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- anlotinib + RAI (Experimental): Patients in this arm will receive anlotinib 6 cycles around RAI treatment ( 4 cycles before and 2 cycles after RAI)
  Interventions: Drug: Anlotinib hydrochloride; Drug: Sodium Iodide I 131
- RAI only (Other): Patients in this arm will receive RAI treatment as scheduled.
  Interventions: Drug: Sodium Iodide I 131
- Penpulimab + RAI (Experimental): Patients in this arm will receive Penpulimab from one week prior to RAI treatment until the disease progressed or intolerable.
  Interventions: Drug: Sodium Iodide I 131; Drug: Penpulimab

INTERVENTIONS:
Drug: Anlotinib hydrochloride — Anlotinib hydrochloride may stop the growth of tumor cells and improve iodine uptake.
  Arms: anlotinib + RAI
Drug: Sodium Iodide I 131 — RAI treatment may shrink the tumor
  Other Names: RAI
Drug: Penpulimab — Penpulimab is a novel structure Immune checkpoint inhibitor. The combination of Penpulimab and RAI might have synergistic effects for DTC.
  Arms: Penpulimab + RAI

SUMMARY:
The purpose of this study is to assess the efficacy and safety of anlotinib in combination with I-131 in locally advanced/metastatic differentiated thyroid cancer. Anlotinib may stop the growth of tumor cells and improve iodine uptake.

DETAILED DESCRIPTION:
Primary Outcome Measures:

objective response rate (ORR)

Secondary Outcome Measures：

1. Biochemical Response Rate (BRR) Biochemical response rate is defined as the percentage of subjects whose Tg was consecutive decreases more than 25% compared to baseline twice
2. Disease Control Rate (DCR)
3. Progression-free Survival (PFS) (median) was determined using the number of months measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression) of participants. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
4. Nuclear medicine functional imaging changes of target lesions The dynamic changes of I uptake and 18F-FDG PET/CT imaging

ELIGIBILITY:
Inclusion Criteria:

* local advanced or metastatic differentiated thyroid cancer (DTC)
* scheduled to receive RAI treatment.
* absence of good remission of RAI or may not get satisfactory remission from RAI treatment
* At least one measurable lesion, with diameter ≥ 10mm measured by spiral MRI/CT scan per RECIST1.1.
* Be 18 years of age or older, ECOG PS: 0-2. Life expectancy of at least 6 months.
* Main organs function is normal.
* The woman patients of childbearing age who must agree to take contraceptive methods (e.g. intrauterine device, contraceptive pill or condom) during the research and within another 6 months after it; who are not in the lactation period and examined as negative in blood serum test or urine pregnancy test within 7 days before the research; The man patients who must agree to take contraceptive methods during the research and within another 6 months after it.

Exclusion Criteria:

* Patients who had previously received treatment with Antiangiogenic tyrosine kinase inhibitors, such as: Anlotinib, apatinib and Lenvatinib.
* Patients who had previously received local treatment within 4 weeks or Participated in other anti-tumor clinical trials within 4 weeks.
* Patients with previous or current concurrent malignancies or solid organs or bone marrow transplants within 5 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Unmitigated ≥ grade 2 toxicity (CTC AE 5.0) due to any prior treatment, excluding alopecia.
* With kinds of factors which affect oral medicine (e.g. failing to swallow, gastrointestinal tract getting resected, chronic diarrhea and ileus)
* Patients with pleural effusion or ascites.
* Patients with any severe and/or uncontrolled disease.
* Patients who underwent major surgery, open biopsy or significant traumatic injury within 4 weeks.
* Regardless of the severity, patients with any physical signs or history of bleeding, patients with bleeding or bleeding events greater than or equal to CTCAE 2 within four weeks prior to the first administration, or patients with unhealed wounds, fractures, ulcers.
* Patients with arterial or venous thromboembolic events occurred within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-07-20 (Estimated); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | up to 24 months
  Proportion of patients with target lesions reaching PR or CR

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | up to 24 months
  Proportion of patients with target lesions reaching PR, CR or SD
Biochemical Response Rate (BRR) | up to 24 months
  Biochemical response rate is defined as the percentage of subjects whose Tg was consecutive decreases more than 25% compared to baseline twice
Progression-free Survival (PFS) (median) | up to 24 months
  PFS was determined using the number of months measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression) of participants. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Nuclear medicine functional imaging changes of target lesions | up to 24 months
  The dynamic changes of I uptake and 18F-FDG PET/CT imaging

CONTACTS AND LOCATIONS:
Overall Officials: Yansong Lin, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No